CLINICAL TRIAL: NCT01100944
Title: A Phase 1/2 Study of PXD101 (Belinostat) in Combination With Cisplatin, Doxorubicin and Cyclophosphamide in the First Line Treatment of Advanced or Recurrent Thymic Malignancies
Brief Title: A Phase 1/2 Study of PXD101 (Belinostat) in Combination With Cisplatin, Doxorubicin and Cyclophosphamide in the First Line Treatment of Advanced or Recurrent Thymic, Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Principal investigator left the National Institutes of Health (NIH).
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100077; 10-C-0077
Record Dates: First submitted 2010-03-18; First posted 2010-04-09 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Thymoma; Thymic Carcinoma
Keywords: Gene Expression; HDAC Class I and II enzymes; Thymoma; Chemotherapy; Hydroxamic Acid Deacetylase Inhibitor; Thymic Cancer
MeSH Terms: conditions — Thymoma; Thymus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Therapy in Thymic Malignancies (Experimental): PXD101 (Belinostat) will be given as a 48h continuous intravenous infusion (CIVI) starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2 and 3, cisplatin will be infused over 1 hour on day 2 and cyclophosphamide as a slow IV infusion on Day 3. Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with PXD101 alone may continue until disease progression. A conventional 3+3 dose escalation design was used with up to 3 additional patients added if one patient exhibited a dose limiting toxicity (DLT). Dose escalation was halted if at least 2 out of a maximum of 6 patients within a cohort exhibited a DLT.
  Interventions: Drug: PXD101with cisplatin+doxorubicin+cyclophosphamide

INTERVENTIONS:
Drug: PXD101with cisplatin+doxorubicin+cyclophosphamide — PXD101 will be given as a 48h continuous intravenous infusion (CIVI) starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2 and 3, cisplatin will be infused over 1 hour on day 2 and cyclophosphamide as a slow IV infusion on Day 3. Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with PXD101 alone may continue until disease progression.

SUMMARY:
Background:

* Tumors of the thymus are rare and can be treated with surgery, but it is often difficult to determine whether a thymic tumor is malignant based on biopsy alone and the long-term survival rate is less than 50 percent. Because thymic tumors are so rare, most treatment knowledge comes from a relatively small series of cases, and the choice of treatment usually depends on the hospital or clinic staff's experience and familiarity with a given chemotherapy and surgery regimen.
* Belinostat is an investigational anticancer drug that has not yet been approved by the Food and Drug Administration for use in any cancer. Researchers are interested in determining whether belinostat can be combined with conventional chemotherapy to safely and effectively treat advanced thymic cancer.

Objectives:

* To determine a safe and tolerable dose of belinostat that can be given in combination with cisplatin, doxorubicin, and cyclophosphamide.
* To determine if belinostat (combined with the abovementioned standard chemotherapy regimen) is effective against thymic cancer cells.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with advanced or recurrent thymic malignancy that is not considered to be curable with surgery or radiation therapy, and who have not received previous chemotherapy treatment.

Design:

* Participants will be screened with a physical exam, blood tests, and imaging studies as directed by the study researchers.
* Participants will receive six 21-day cycles (18 weeks) of treatment with belinostat in combination with cisplatin, doxorubicin, and cyclophosphamide. The treatment will require continuous infusion over 3 days, and participants will remain in the treatment center during this time. Participants will have regular blood tests, clinic visits, and imaging studies during the treatment period.
* Participants who complete the six treatment cycles with no severe side effects may be offered the option to continue treatment with belinostat alone.
* After the 18-week study period, participants will return for regular follow-up exams for at least 4 weeks, and will be asked to remain in contact with the study researchers once a year to continue to study long-term effects....

DETAILED DESCRIPTION:
Background:

* New options for the treatment of patients with advanced thymoma and thymic carcinoma are needed.
* Belinostat, N-hydroxy-3-(phenylsulphamoylphenyl) acrylamide, is a hydroxamic acid deacetylase inhibitor that is able to inhibit both histone deacetylase inhibitors (HDAC) Class I and II enzymes.
* An ongoing phase II study of belinostat in recurrent or metastatic thymic malignancies has shown activity which warrants further consideration of belinostat in the first line.
* Belinostat alterations in target protein levels due to gene expression changes may allow increased sensitivity of cancer cells to conventional chemotherapy.

Objectives:

Primary Objectives

* In the Phase I portion the primary objective will be to determine a safe and tolerable phase 2 dose, dose limiting toxicities (DLTs) and preliminary activity for the combination of belinostat by continuous intravenous (IV) infusion (CIVI) with cisplatin, doxorubicin and cyclophosphamide in patients with advanced thymic malignancies.
* In the Phase II portion the primary objective will be to determine the clinical response rate (partial response (PR)+complete response (CR)) of belinostat in combination with cisplatin, doxorubicin and cyclophosphamide in the first line treatment of patients with advanced thymic malignancies.

Secondary Objectives

* To determine time to response, duration of response, progression free survival (PFS) and overall survival (OS).
* To determine the toxicity profile and safety of this combination.
* To assess exploratory correlative markers in relation to response to treatment (immunohistochemistry and array Comparative Genomic Hybridization (CGH))

Eligibility:

* Patients with histologically confirmed advanced thymic malignancies who are chemotherapy na(SqrRoot) ve.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Adequate renal, hepatic and hematopoietic function

Design:

* The Phase I portion of the study will consist of four dose levels and dose escalations will follow according to traditional 3 patient cohorts.
* Once the maximum tolerated doe is determined, the phase II portion of the study will begin.
* Belinostat will be given as a 48h CIVI starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2 and 3, cisplatin will be infused over 1 hour on day 2 and cyclophosphamide as a slow IV infusion on Day 3.
* Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with belinostat alone may continue until disease progression.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Both the phase I and phase II portions of the protocol will be only open to patients with histologically confirmed advanced stage (Masaoka stage III or IV) thymic malignancies.
2. Patients must be chemotherapy na(SqrRoot) ve for the treatment of advanced thymic malignancies.
3. Age > 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%).
5. Life expectancy of greater than 3 months.
6. Patients must have normal organ and marrow function as defined below:

   * leukocytes > 3,000/mcL
   * absolute neutrophil count > 1,500/mcL
   * platelets > 100,000/mcL
   * total bilirubin within normal institutional limits
   * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 5 times the institutional upper limit of normal with evidence of metastatic disease to the liver or less than or equal to 3 times the institutional upper limit of normal without evidence of metastatic disease to the liver
   * creatinine less than or equal to 1.5 times institutional upper limits of normal

   OR

   - creatinine clearance > 45 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
7. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan.
8. Patients must have recovered from toxicity related to prior therapy (surgery or radiation) to grade less than or equal to 1 and must be at least 28 days since any prior radiation or major surgery.

   Target lesions cannot be selected within previously irradiated areas, if not newly arising or clearly progressing after irradiation as proven by repeat scanning.
9. Concurrent corticosteroids for myasthenia gravis, or other paraneoplastic syndromes, or other chronic conditions are allowed.

   Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of belinostat or cisplatin, doxorubicin or cyclophosphamide will be determined following review of their case by the Principal Investigator. Efforts should be made to switch patients with brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications.
10. The effects of belinostat on the developing human fetus are unknown. For this reason and because histone deacetylase inhibitors (HDAC) inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. Ability to understand and the willingness to sign a written informed consent document.

Inclusion of Women and Minorities

Both men and women of all races and ethnic groups are eligible for this trial

EXCLUSION CRITERIA:

1. Patients who have had major surgery or radiotherapy within 3 weeks of enrollment.
2. Patients may not be receiving any other investigational agents.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 1 month without steroids may be enrolled at the discretion of the principal investigator.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to belinostat or other agents used in study.
5. Patients with prior treatment with drugs of the HDAC inhibitor class are excluded, except for valproic acid (VPA) where prior treatment is accepted as long as it is not within the last 2 weeks before enrolment.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because belinostat is an HDAC inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with belinostat, breastfeeding should be discontinued if the mother is treated with belinostat. These potential risks may also apply to other agents used in this study.
8. Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with belinostat. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
9. Marked baseline prolongation of Q wave, T wave (QT)/corrected QT interval (QTc) interval, e.g., repeated demonstration of a QTc interval > 500 ms; Long QT Syndrome. Patients taking medications that may cause QTc prolongation will be eligible as long as they comply with the recommendations in appendix D.
10. History of another invasive malignancy in the last five years. Adequately treated non-invasive, non-melanoma skin cancers as well as in situ carcinoma of the cervix will be allowed.
11. Patients with tumor amenable to potentially curative therapy as assessed by the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2015-10-21 (Actual); Study Completion 2015-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girard N, Mornex F, Van Houtte P, Cordier JF, van Schil P. Thymoma: a focus on current therapeutic management. J Thorac Oncol. 2009 Jan;4(1):119-26. doi: 10.1097/JTO.0b013e31818e105c. PMID 19096319
- [Background] Loehrer PJ Sr, Kim K, Aisner SC, Livingston R, Einhorn LH, Johnson D, Blum R. Cisplatin plus doxorubicin plus cyclophosphamide in metastatic or recurrent thymoma: final results of an intergroup trial. The Eastern Cooperative Oncology Group, Southwest Oncology Group, and Southeastern Cancer Study Group. J Clin Oncol. 1994 Jun;12(6):1164-8. doi: 10.1200/JCO.1994.12.6.1164. PMID 8201378
- [Background] Giaccone G. Treatment of malignant thymoma. Curr Opin Oncol. 2005 Mar;17(2):140-6. doi: 10.1097/01.cco.0000152628.43867.8e. PMID 15725919
- [Result] Thomas A, Rajan A, Szabo E, Tomita Y, Carter CA, Scepura B, Lopez-Chavez A, Lee MJ, Redon CE, Frosch A, Peer CJ, Chen Y, Piekarz R, Steinberg SM, Trepel JB, Figg WD, Schrump DS, Giaccone G. A phase I/II trial of belinostat in combination with cisplatin, doxorubicin, and cyclophosphamide in thymic epithelial tumors: a clinical and translational study. Clin Cancer Res. 2014 Nov 1;20(21):5392-402. doi: 10.1158/1078-0432.CCR-14-0968. Epub 2014 Sep 4. PMID 25189481
- [Derived] Giaccone G, Rajan A, Berman A, Kelly RJ, Szabo E, Lopez-Chavez A, Trepel J, Lee MJ, Cao L, Espinoza-Delgado I, Spittler J, Loehrer PJ Sr. Phase II study of belinostat in patients with recurrent or refractory advanced thymic epithelial tumors. J Clin Oncol. 2011 May 20;29(15):2052-9. doi: 10.1200/JCO.2010.32.4467. Epub 2011 Apr 18. PMID 21502553
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0077.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Belinostat 250mg/m(2) and Chemotherapy: Patients received 250mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
- Belinostat 500mg/m(2) and Chemotherapy: Patients received 500mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
- Belinostat and Chemotherapy at the Maximum Tolerated Dose(MTD): Patients were treated with belinostat, doxorubicin, cisplatin and cyclophosphamide at the maximum tolerated dose derived from the phase I dose level.
Period: Dose Escalation Phase 1 Dose Level 1
Arm/Group | Belinostat 250mg/m(2) and Chemotherapy | Belinostat 500mg/m(2) and Chemotherapy | Belinostat and Chemotherapy at the Maximum Tolerated Dose(MTD)
Started | 6 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Discontinued due to treatment delay | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Period: Dose Escalation Phase 1 Dose Level 2
Arm/Group | Belinostat 250mg/m(2) and Chemotherapy | Belinostat 500mg/m(2) and Chemotherapy | Belinostat and Chemotherapy at the Maximum Tolerated Dose(MTD)
Started | 0 | 2 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Period: Expansion Phase - Phase 2
Arm/Group | Belinostat 250mg/m(2) and Chemotherapy | Belinostat 500mg/m(2) and Chemotherapy | Belinostat and Chemotherapy at the Maximum Tolerated Dose(MTD)
Started | 0 | 0 | 18
Completed | 0 | 0 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol, two group results, as well as single arm results are reported throughout the results data.
Groups:
- All Participants: All participants who had at least one dose of Belinostat.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG).
  Grade 0 is normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    Grade 0 | 18
    Grade 1 | 8
Tumor Type [Count of Participants; unit: Participants] — The World Health Organization (WHO) classification of epithelial thymic malignancies shown under Thymoma are defined as type B1: histology - predominantly cortical thymoma, type B2: histology - cortical thymoma, and type B3: histology - well-differentiated thymoma.
  Participants
    Thymoma | 12
    B1 | 2
    B2 | 7
    B3 | 3
    Thymic carcinoma | 14
Stage at Enrolment [Count of Participants; unit: Participants] — Masaoka Staging System:
  Stage IVA is pleural or pericardial dissemination. Stage IVB is lymphogenous or hematogenous metastases.
  Participants
    IVA | 12
    IVB | 14
Prior Surgery [Count of Participants; unit: Participants] — 11 patients had radical surgery including 2 who underwent debulking subsequently.
  Participants
    Radical | 11
    Debulking | 2
Prior Radiation [Count of Participants; unit: Participants] | 7
Prior Neoadjuvant or Adjuvant Chemotherapy [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Belinostat
Description: The MTD is defined as the highest dose at which less than 2 out of 6 patients experienced a dose limiting toxicity (DLT). A DLT is defined as grade 4 neutropenia lasting more than 7 days despite prophylactic or therapeutic use of granulocyte colony-stimulating factor (G-CSF), febrile neutropenia defined as absolute neutrophil count (ANC) less than 1000/mm(3) and temperature more than 38.5 degrees Celsius or 100.4 degrees Fahrenheit or life threatening sepsis, grade 4 thrombocytopenia or grade 3 thrombocytopenia associated with bleeding during the first cycle of therapy. Any grade 3 or 4 non-hematologic toxicity was considered dose limiting with the following exceptions: grade 3 diarrhea lasting less than 48 hours, grade 3 nausea and/or vomiting lasting less than 48 hours, grade 3 electrolyte abnormalities lasting less than 48 hours, grade 3 creatinine elevation lasting less than 48 hours.
Time Frame: 2 years
Measure: Number; unit: mg/m(2)
Groups:
- Phase I Dose Level 1 & Phase I Dose Level 2: Patients received 250mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
Arm/Group | Phase I Dose Level 1 & Phase I Dose Level 2
Number analyzed (Participants) | 8
mg/m(2) | 1000

2. Primary Outcome: Number of Participants With Grade 3 and 4 Dose Limiting Toxicity (DLT) at 2000mg/m(2) Belinostat
Description: A DLT is defined as grade 4 neutropenia lasting more than 7 days despite prophylactic or therapeutic use of granulocyte colony-stimulating factor (G-CSF), febrile neutropenia defined as absolute neutrophil count (ANC) less than 1000/mm(3) and temperature more than 38.5 degrees Celsius or 100.4 degrees Fahrenheit or life threatening sepsis, grade 4 thrombocytopenia or grade 3 thrombocytopenia associated with bleeding during the first cycle of therapy. Any grade 3 or 4 non-hematologic toxicity was considered dose limiting with the following exceptions: grade 3 diarrhea lasting less than 48 hours, grade 3 nausea and/or vomiting lasting less than 48 hours, grade 3 electrolyte abnormalities lasting less than 48 hours, grade 3 creatinine elevation lasting less than 48 hours.
Time Frame: up to 122 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Level 2: Patients received 500mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
Arm/Group | Phase I Dose Level 2
Number analyzed (Participants) | 2
Participants
  Grade 3 Nausea | 2
  Grade 3 Diarrhea | 2
  Grade 4 Neutropenia | 2
  Grade 4 Thrombocytopenia | 2

3. Primary Outcome: Objective Response Rate (Partial Response (PR) + Complete Response (CR) of Belinostat in Combination With Cisplatin, Doxorubicin and Cyclophosphamide in the First Line Treatment of Patients With Advanced Thymic Malignancies
Description: Objective response rate is the number of participants with a best objective response of partial response (PR) + complete response (CR) per the Response Criteria in Solid Tumors (RECIST) divided by the number of participants who had treatment.
Time Frame: 43 months
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Thymic Participants; Thymoma Participants: The thymic tumors are rare tumors that arise from the thymus and are histologically composed of epithelial cells which are the putative source of malignancy, B and T lymphocytes, interdigitating reticulum cells, macrophages, and myeloid cells. The most common tumors of the thymus are thymomas (well-differentiated neoplasms), atypical thymomas (moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
- Thymic and Thymoma Participants: All participants who had at least one dose of belinostat. PXD101 (Belinostat) will be given as a 48h continuous intravenous infusion (CIVI) starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2, 3, cisplatin will be infused over 1 hr on day 2 and cyclophosphamide as a slow IV infusion on Day 3. Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with PXD101 alone may continue until disease progression.
  The thymic tumors are rare tumors that arise from the thymus and are histologically composed of epithelial cells which are the putative source of malignancy, B and T lymphocytes, interdigitating reticulum cells, macrophages, and myeloid cells. The most common tumors of the thymus are thymomas (well-differentiated neoplasms), atypical thymomas (moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
Arm/Group | Thymic Participants | Thymoma Participants | Thymic and Thymoma Participants
Number analyzed (Participants) | 14 | 11 | 25
percentage of participants | 21 [4.7 to 50.8] | 64 [30.8 to 89.1] | 40 [21.1 to 61.3]

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events. For a detailed list of events, see the adverse event module.
Time Frame: up to 122 months
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who had at least one dose of belinostat. PXD101 (Belinostat) will be given as a 48h continuous intravenous infusion (CIVI) starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2, 3, cisplatin will be infused over 1 hr on day 2 and cyclophosphamide as a slow IV infusion on Day 3. Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with PXD101 alone may continue until disease progression.
  The thymic tumors are rare tumors that arise from the thymus and are histologically composed of epithelial cells which are the putative source of malignancy, B and T lymphocytes, interdigitating reticulum cells, macrophages, and myeloid cells. The most common tumors of the thymus are thymomas (well-differentiated neoplasms), atypical thymomas (moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Participants
  Serious | 20
  Non-serious | 26

5. Secondary Outcome: Treatment-related Grade 3 and 4 Adverse Events (Highest Grade Per Event Per Patient)
Description: Here are the number of patients with treatment -related grade 3 and 4 adverse events (highest grade per event per patient).
Time Frame: up to 122 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Level 1 + Phase 2: Patients received 250mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD) and was utilized in the expansion phase (phase 2).
Arm/Group | Phase I Dose Level 1 + Phase 2 | Phase I Dose Level 2 | All Participants
Number analyzed (Participants) | 24 | 2 | 26
Participants
  Hematologic: Lymphocyte count decreased | 24 | 2 | 26
  Hematologic: White blood cell decreased | 22 | 2 | 24
  Hematologic: Neutrophil count decreased | 19 | 2 | 21
  Hematologic: Platelet count decreased | 10 | 2 | 12
  Hematologic: Anemia | 7 | 2 | 9
  Hepatic and Renal: Hypophosphatemia | 4 | 2 | 6
  Hepatic and Renal: Aspartate aminotransferase incr | 4 | 2 | 6
  Hepatic/Renal: Alanine aminotransferase increased | 3 | 1 | 4
  Hepatic and Renal: Hypokalemia | 3 | 1 | 4
  Hepatic and Renal: Hypermagnesemia | 3 | 0 | 3
  Hepatic and Renal: Hypoalbuminemia | 1 | 1 | 2
  Hepatic and Renal: Hypocalcemia | 1 | 1 | 2
  Hepatic and Renal: Hypomagnesemia | 1 | 0 | 1
  Hepatic and Renal: Hyponatremia | 1 | 0 | 1
  Cardiovascular: Thromboembolic event | 3 | 0 | 3
  Cardiovascular: Atrial fibrillation | 0 | 1 | 1
  Cardiovascular: Ejection fraction decreased | 1 | 0 | 1
  Cardiovascular: Electrocardiogram QTc prolonged | 1 | 0 | 1
  Others: Nausea | 1 | 2 | 3
  Other: Febrile neutropenia | 3 | 0 | 3
  Others: Diarrhea | 1 | 1 | 2
  Others: Lung infection | 2 | 0 | 2
  Otehrs: Entercolitis infectious | 1 | 1 | 2
  Others: Fatigue | 2 | 0 | 2
  Others: Hearing impaired | 1 | 0 | 1
  Others: Hypoxia | 1 | 0 | 1
  Others: Non-cardiac chest pain | 1 | 0 | 1
  Others: Pain in extremity | 1 | 0 | 1
  Others: Syncope | 1 | 0 | 1
  Others: Tumor lysis syndrome | 0 | 1 | 1
  Others: Limb edema | 0 | 1 | 1
  Others: Urinary tract infection | 1 | 0 | 1
  Others: Vomiting | 0 | 1 | 1

6. Secondary Outcome: Clinical Response
Description: Response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 43 months
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable for response.
Measure: Count of Participants; unit: Participants
Groups:
- Thymic Particpants; Thymoma Participants: PXD101 (Belinostat) will be given as a 48h continuous intravenous infusion (CIVI) starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2, 3, cisplatin will be infused over 1 hr on day 2 and cyclophosphamide as a slow IV infusion on Day 3. Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with PXD101 alone may continue until disease progression.
  The thymic tumors are rare tumors that arise from the thymus and are histologically composed of epithelial cells which are the putative source of malignancy, B and T lymphocytes, interdigitating reticulum cells, macrophages, and myeloid cells. The most common tumors of the thymus are thymomas (well-differentiated neoplasms), atypical thymomas (moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
Arm/Group | Thymic Particpants | Thymoma Participants | Thymic and Thymoma Participants
Number analyzed (Participants) | 14 | 11 | 25
Participants
  Complete Response (CR) | 0 | 1 | 1
  Partial Response (PR) | 3 | 6 | 9
  Stable Disease (SD) | 10 | 4 | 14
  Progressive Disease (PD) | 1 | 0 | 1

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as stable disease (SD) + partial response (PR) + complete response (CR) per the Response Criteria in Solid Tumors (RECIST).
Time Frame: 43 months
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Thymic Participants; Thymoma Participants: PXD101 (Belinostat) will be given as a 48h continuous intravenous infusion (CIVI) starting on day 1, doxorubicin as a slow intravenous (IV) injection on days 2, 3, cisplatin will be infused over 1 hr on day 2 and cyclophosphamide as a slow IV infusion on Day 3. Treatment will be given every 21 days for no more than 6 cycles or until disease progression. Treatment with PXD101 alone may continue until disease progression.
  The thymic tumors are rare tumors that arise from the thymus and are histologically composed of epithelial cells which are the putative source of malignancy, B and T lymphocytes, interdigitating reticulum cells, macrophages, and myeloid cells. The most common tumors of the thymus are thymomas (well-differentiated neoplasms), atypical thymomas (moderately differentiated neoplasms) and thymic (poorly differentiated neoplasms) carcinomas.
Arm/Group | Thymic Participants | Thymoma Participants | Thymic and Thymoma Participants
Number analyzed (Participants) | 14 | 11 | 25
percentage of participants | 93 [66.1 to 99.8] | 100 [71.5 to 100] | 96 [79.7 to 99.9]

8. Secondary Outcome: Time to Response
Description: Time to response is the time between the first day of treatment until first date of response (complete response (CR) + partial response (PR)) (whichever is first recorded).
Time Frame: From the first day of treatment until the date of first documented response, assessed up to 43 months
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable for response.
Measure: Median (Full Range); unit: days
Groups:
- Phase I Dose Level 1 & Phase I Dose Level 2: Patients received 250mg/m(2) or 500mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
Arm/Group | Phase I Dose Level 1 & Phase I Dose Level 2
Number analyzed (Participants) | 25
days | 44.5 [39 to 110]

9. Secondary Outcome: Duration of Response
Description: Duration of response is measured from the time measurement criteria (e.g. Response Evaluation Criteria in Solid Tumors (RECIST)) are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: From the time of first response until date of progression, assessed up to 43 months
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable for response. The reason median was not reached is that patients with thymoma have a more indolent disease with a longer survival, therefore a longer duration of response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thymic Participants | Thymoma Participants | Thymic and Thymoma Participants
Number analyzed (Participants) | 14 | 11 | 25
months | 7.4 [4.2 to 8.5] | NA [NA to NA] — Median duration of response was not reached for thymoma participants. | 7.4 [5.2 to NA] — 5.2 months to undefined upper limit.

10. Secondary Outcome: Progression Free Survival (PFS)
Description: Duration of time from start of treatment to time of progression or death whichever occurs first.
Time Frame: Start of treatment to time of disease progression or death whichever occurs first, assessed up to 43 months
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable. The reason median was not reached is that patients with thymoma have a more indolent disease with a longer survival, therefore a longer duration of response.
Measure: Median (Full Range); unit: months
Arm/Group | Thymic Participants | Thymoma Participants | Thymic and Thymoma Participants
Number analyzed (Participants) | 14 | 11 | 25
months | 7.2 [2 to 9] | NA [5 to 32] — Median PFS was not reached for thymoma participants. | 9 [2 to 32]
Statistical Analysis 1: Comparison: Thymic and Thymoma Participants; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the on-study date until the date of death or progression as appropriate.
Time Frame: Start of treatment to time of death, assessed up to 43 months
Population: as for outcome 10
Measure: Median (Full Range); unit: months
Arm/Group | Thymic Participants | Thymoma Participants | Thymic and Thymoma Participants
Number analyzed (Participants) | 14 | 11 | 25
months | 21.4 [3 to 37] | NA [4 to 43] — Median OS was not reached for thymoma participants. Thymoma patients with maximum and minimum OS values were alive at the time of data cutoff. | 28.5 [3 to 43]

12. Secondary Outcome: Time to Half Life (t1/2) of Belinostat
Description: Half life is the duration of time for the drug to be reduced to half the original amount.
Time Frame: on day 1: pre-belinostat and 0, 0.5, 1 and 2 hours after belinostat infusion, on day 3: 0, 0.8, 0.25, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-last belinostat dose.
Measure: Mean (Standard Deviation); unit: Hour
Groups:
- Phase 1 Dose Level 1 + Phase 2: Patients received 250mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
- Phase 1 Dose Level 2: Patients received 500mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
Arm/Group | Phase 1 Dose Level 1 + Phase 2 | Phase 1 Dose Level 2
Number analyzed (Participants) | 24 | 1
Hour | 0.47 (0.19) | 0.40 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

13. Secondary Outcome: Total Clearance (CL) of Belinostat
Description: Clearance is the amount of time for the drug to be eliminated from the body.
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Phase 1 Dose Level 1 + Phase 2 | Phase 1 Dose Level 2
Number analyzed (Participants) | 24 | 1
L/hr | 133.5 (145.1) | 132.1 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Belinostat
Description: Plasma concentrations of Belinostat were measured using a newly designed and validated ultra high-performance liquid chromatography (HPLC) with tandem mass spectrometric (MS/MS) assay, with a lower limit of quantification of 5ng/mL.
Time Frame: as for outcome 12
Population: One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2. Dose normalized parameters are normalized to absolute total dose (over 48 hours continuous intravenous infusion (CIVI)) for that patient, not dose level.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Phase I Dose Level 1 + Phase 2: Patients received 250mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
Arm/Group | Phase I Dose Level 1 + Phase 2 | Phase I Dose Level 2
Number analyzed (Participants) | 24 | 1
ng/ml | 650.6 (288.1) | 1202 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

15. Secondary Outcome: Maximum Plasma Concentration (Cmax)/Dose
Description: as for outcome 14
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml/mg
Arm/Group | Phase I Dose Level 1 + Phase 2 | Phase I Dose Level 2
Number analyzed (Participants) | 24 | 1
ng/ml/mg | 0.36 (0.21) | 0.31 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

16. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to reach peak concentration after drug administration.
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Phase I Dose Level 1 + Phase 2 | Phase I Dose Level 2
Number analyzed (Participants) | 24 | 1
Hour | 25.28 (22.29) | 50.0 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

17. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve Extrapolated to Infinity (AUC(INF))
Description: AUC is a measure of the serum concentration of Belinostat over time. It is used to characterize drug absorption.
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Phase I Dose Level 1 + Phase 2 | Phase I Dose Level 2
Number analyzed (Participants) | 24 | 1
hr*ng/ml | 19756 (7634) | 29686 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

18. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve Extrapolated to Infinity (AUC(INF)/Dose
Description: AUC is a measure of the serum concentration of Belinostat over time. It is used to characterize drug absorption.
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr*ng/ml/mg
Arm/Group | Phase I Dose Level 1 + Phase 2 | Phase I Dose Level 2
Number analyzed (Participants) | 24 | 1
hr*ng/ml/mg | 10.78 (5.57) | 7.57 (NA) — One patient was excluded from pharmacokinetic analysis due to insufficient sampling in dose level 2.

19. Secondary Outcome: Relative Change Observed in Total Protein Hyperacetylation of Cluster of Differentiation 3 (CD3)+T Cells With Belinostat
Description: Changes in marker levels from baseline. All pre values were set to 1 so that we could measure changes relative to the baseline.
Time Frame: Baseline Cycle 1 Day 1 (C1D1), Cycle 1 Day 2 (C1D2), Cycle 1 Day 3 (C1D3), and Cycle 2 Day 1 (C2D1)
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable. Two samples could not be analyzed since they were of poor quality with too few cells for immune cell subset analysis or the samples could not be collected in time for pharmacodynamics analysis.
Measure: Median (Full Range); unit: Relative fold change
Groups:
- All Participants: Patients received 250mg/m(2) or 500mg/m(2) of belinostat via four consecutive 12 hour continuous intravenous infusion (CIVI) for 48 hours starting on day 1. At dose levels 1 and 2, patients received the same doses of doxorubicin (25mg/m(2) on days 2 and 3, intravenous push over 3-5 minutes), cisplatin (50 mg/m(2) over 60 minutes intravenous on day 2 after doxorubicin), and cyclophosphamide (500mg/m(2) over 60 minutes intravenous on day 3 after doxorubicin). Combination of chemotherapy and belinostat was repeated every 21 days for a total of 6 cycles unless there was evidence of disease progression or intolerance of the study treatment.
  A conventional 3 + 3 dose escalation design was used to determine maximum tolerated dose (MTD).
Arm/Group | All Participants
Number analyzed (Participants) | 23
Relative fold change
  C1D2 | 3.45 [0.96 to 14.29]
  C1D3 | 2.49 [0.98 to 10.74]
  C2D1 | 1.15 [0.97 to 2.40]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.30, Wilcoxon signed rank test — Fold change at Cycle 2 Day 1 vs. pre was assessed. Only differences with p<0.005 could be potentially considered statistically significant while those with 0.005<p<0.05 would represent trends towards a difference
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test — Fold change at Cycle 1 Day 2 vs. pre was assessed. p values calculated were done using a Wilcoxon signed rank test relative to a ratio of 1
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test — Fold change at Cycle 1 Day 3 vs. pre was assessed. p values calculated were done using a Wilcoxon signed rank test relative to a ratio of 1

20. Secondary Outcome: Relative Changes in the Number of Tregs With Treatment
Description: as for outcome 19
Time Frame: Baseline Cycle 1 Day 1 (C1D1), Cycle 1 Day 2 (C1D2), Cycle 1 Day 3 (C1D3), and Cycle 2 Day 1 (C2D1)
Population: One patient hospitalized for viral meningoencephalitis during the first cycle was not evaluable. Three samples could not be analyzed since they were of poor quality with too few cells for immune cell subset analysis or the samples could not be collected in time for pharmacodynamics analysis.
Measure: Median (Full Range); unit: relative fold change
Arm/Group | All Participants
Number analyzed (Participants) | 22
relative fold change
  C1D2 | 0.58 [0.03 to 1.88]
  C1D3 | 0.47 [0 to 1.58]
  C2D1 | 1.12 [0.12 to 2.55]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.76, Wilcoxon signed rank test — Fold change at Cycle 2 Day 1 vs. pre was assessed.Only differences with p<0.005 could be potentially considered statistically significant while those with 0.005<p<0.05 would represent trends towards a difference
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; p = 0.0009, Wilcoxon signed rank test — [p-value comment as in outcome 19, analysis 2]
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 19, analysis 3]

21. Secondary Outcome: Relative Changes in T Cell Immunoglobulin Domain and Mucin Domain-3 (TIM3)-Expressing Cluster of Differentiation 8 (CD8)+Tcells
Description: as for outcome 19
Time Frame: Baseline Cycle 1 Day 1 (C1D1), Cycle 1 Day 2 (C1D2), Cycle 1 Day 3 (C1D3), and Cycle 2 Day 1 (C2D1)
Population: as for outcome 20
Measure: Median (Full Range); unit: Relative fold change
Arm/Group | All Participants
Number analyzed (Participants) | 22
Relative fold change
  C1D2 | 0.81 [0.57 to 1.25]
  C1D3 | 0.66 [0.42 to 0.91]
  C2D1 | 1.01 [0.67 to 1.31]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.95, Wilcoxon signed rank test — Fold change at Cycle 2 Day 1 vs. pre was assessed. p values calculated were done using a Wilcoxon signed rank test relative to a ratio of 1
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 19, analysis 2]
Statistical Analysis 3: Comparison: All Participants; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test — [p-value comment as in outcome 19, analysis 3]

ADVERSE EVENTS:
Time Frame: up to 122 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 13/26
Serious Adverse Events (participants affected / at risk) | 20/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=26)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2)
Death NOS (General disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations - Other, Meningoencephylitis (Infections and infestations) | 1 (1)
Infections and infestations - Other, West Nile virus (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other,Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=26)
Activated partial thromboplastin time prolonged (Investigations) | 3 (6)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (26)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 23 (124)
Anorexia (Metabolism and nutrition disorders) | 15 (18)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 10 (25)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chills (General disorders) | 3 (3)
Concentration impairment (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Creatinine increased (Investigations) | 4 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 9 (18)
Dizziness (Nervous system disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Edema limbs (General disorders) | 4 (5)
Ejection fraction decreased (Investigations) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 8 (27)
Enterocolitis infectious (Gastrointestinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 15 (28)
Fever (General disorders) | 3 (3)
Floaters (Eye disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Hearing impaired (Ear and labyrinth disorders) | 2 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (7)
Hypertension (Vascular disorders) | 3 (52)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (66)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (58)
Hypokalemia (Metabolism and nutrition disorders) | 7 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (14)
Hyponatremia (Metabolism and nutrition disorders) | 3 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (34)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Infections and infestations - Other, folliculitis, axilla right (Infections and infestations) | 1 (1)
Infections and infestations - Other, Pseudomonas bacteremia (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Laryngitis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 26 (294)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (8)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 16 (21)
Neutrophil count decreased (Investigations) | 24 (112)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Pain (General disorders) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Pharyngitis (Infections and infestations) | 3 (4)
Platelet count decreased (Investigations) | 17 (82)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Presyncope (Nervous system disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (6)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Sinusitis (Infections and infestations) | 3 (3)
Skin and subcutaneous tissue disorders - Other, Basal Cell Carcinoma per biopsy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Ecchymotic nod L arm (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 3 (5)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (10)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 26 (161)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No